CLINICAL TRIAL: NCT05335395
Title: SUNRISE Cluster RCT: Scaling Up Nurturing Care, a Radio Intervention to Stimulate Early Child Development in Burkina Faso
Brief Title: SUNRISE CRT: Radio Intervention to Stimulate Early Child Development
Acronym: SUNRISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Wellcome Trust (Other); National Institute for Health Research, United Kingdom (Other Government); Development Media International (Other); University College, London (Other); Innovations for Poverty Action (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EPPHZS42
Record Dates: First submitted 2022-04-01; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Child Development

STUDY DESIGN:
Intervention Model Description: This a cluster RCT. Local radio stations in the 8 intervention clusters will broadcast the SUNRISE campaign which will be promoting responsive caregiving and providing opportunities for early learning to support child development during the first 3 years of life. Radio stations in the 7 control clusters will broadcast as normal.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Although the nature of the intervention precludes formal masking of fieldworkers during data collection, we believe that this is unlikely to lead to bias for the following reasons: the data collection will be carried out completely independently of the campaign team; emphasis throughout training will be on understanding early child development, rather than on evaluating the radio campaign; the assessments will follow standardized data collection protocols; and the coders of the responsive parenting videos will be blind to their allocation status. In addition, the strict "blinding" procedures for data analysis described above have been designed to avoid any bias in methodological decisions or interpretation of findings all analyses will first be conducted blind to intervention allocation as. Finally, the randomisation was carried out and the code held by the independent trial statistician; it will only be shared with the campaign team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SUNRISE clusters (Experimental): SUNRISE campaign broadcast through local radio stations plus broadcasting as usual
  Interventions: Behavioral: SUNRISE radio campaign
- Control clusters (No Intervention): Local radio stations broadcast as usual

INTERVENTIONS:
Behavioral: SUNRISE radio campaign — The SUNRISE radio campaign will be promoting responsive caregiving and providing opportunities for early learning to support child development during the first 3 years of life.
  The SUNRISE campaign will follow DMI's established intervention approach with:
  1. 60-second radio spots, tailored to increase awareness, knowledge, motivation, skills and opportunity regarding the target behaviours, will include scripted dramas and modelling of responsive parent-child interactions. Each spot will be broadcast 10 times a day for a week; the content of the spots will be changed on a weekly basis. This weekly cycle will continue for three years.
  2. Long format 60-minute programmes broadcast 2-3 times a week, incorporating longer dramas, real life testimonials and practical 'how to' advice, with space for listeners to call in, express opinions and uncertainties and ask questions.
  Arms: SUNRISE clusters

SUMMARY:
SUNRISE aims to develop and evaluate a radio campaign to promote nurturing care behaviours in the first 3 years of life, particularly responsive parenting and providing opportunities for early learning. The campaign will be broadcast by local radio stations in Burkina Faso for 3 years and comprise: 60-second radio 'spots' including scripted dramas and modelling of responsive parent-child interactions, broadcast 10 times a day in weekly cycles; plus long format evening programs 2-3 times/week, incorporating longer dramas, real life testimonials and practical 'how to' advice, with space for listeners to call in, express opinions and ask questions. The campaign's impact on early child development (ECD) will be evaluated using a cluster RCT design, alongside a process and health economic evaluation.

DETAILED DESCRIPTION:
STUDY AIMS

SUNRISE aims to develop and evaluate, in a cluster randomised trial, a radio campaign in Burkina Faso, to promote nurturing care behaviours in the first 3 years of life, focusing particularly on responsive parenting and providing opportunities for early learning. Children's developmental outcomes will be assessed over the lifetime of the intervention until children are aged 30-32 months.

TRIAL CLUSTERS The trial clusters are defined by the broadcast reach of local radio stations. Eligible clusters for the trial were identified as follows. First 23 potential clusters in areas of Burkina Faso where there is no security risk were identified by modelling the reach and signal strength of local radio stations based on tower location, antenna characteristics, and terrain features. A media survey was then carried out to check the radio stations listened to in each of these clusters. This resulted in 15 clusters which satisfy the following conditions: there are at most two dominant radio stations within the cluster; there is no discernible broadcast from stations in neighbouring clusters; they are not based in the large cities of Ouagadougou or Bobo-Dioulassou; and they are not subject to any security risk.

MAPPING EVALUATION AREAS (EAs) Trial participants will be recruited from an evaluation area within each cluster that is close to the radio station(s), has a high signal strength confirmed by a motorbike survey and likely to have a high listenership based on the media survey. The following will be excluded from the area: towns, villages within 5 Km of towns, villages already on the national electricity grid and villages with populations of 5000 or more as they are likely to be a priority for the national electrification programme.

BASELINE SURVEY

DATA COLLECTION

A baseline survey was carried out before the start of the campaign. Participants were all eligible mothers with a child/children aged less than 3 years. Data comprised socio-demographic and socio-economic factors; parental education levels and literacy; and radio ownership and listening patterns. In addition, the fieldworkers administered the following to mothers of children aged 2 years:

* The short form of the Caregiver Reported Early Development Instruments (CREDI) which is designed to serve as a population-level measure of ECD for children from birth to age three, and which has 20 questions primarily focused on milestones and behaviours that are easy for caregivers to understand, observe, and describe.
* Questions from the support for learning/stimulating environment section of the Family Care Indicators (FCI) survey developed by UNICEF to assess key caregiving/family home environment variables considered critical for early child development. This has been used very extensively, including in the global MICS surveys.

Data from the baseline was used to:

1. Inform the content of the SUNRISE radio campaign.
2. Provide a sampling frame for the surveillance system of 3-monthly household visits that will be used to recruit trial participants and conduct ECD assessments with GIS maps of households within the EAs.
3. Carry out the restricted randomization (see section below).

RANDOMISATION OF CLUSTERS

The SUNRISE campaign will be broadcast by the local radio stations in eight of the clusters chosen at random to be in the intervention group; the other 7 clusters will be in the control group and their radio stations will continue to broadcast as normal. This was carried out using restricted randomization to ensure that the intervention and control clusters were balanced at baseline with respect to radio exposure and predictors of ECD outcomes as follows:

Mean CREDI z-score; difference between intervention and control groups to be a maximum of 0.1.

Mean % key FCI behaviours followed by mothers; difference between intervention and control groups to be a maximum of 10%.

* mothers listening to the radio in the last week; difference between intervention and control groups to be a maximum of 10%.
* mothers who are literate; difference between intervention and control groups to be a maximum of 10%.

The restricted randomization was carried out by the independent trial statistician using the cvcrand command in Stata. This performs covariate-constrained randomisation which is suitable for cluster randomised trials with a small number of clusters.

PARTICIPANTS At least 125 eligible children born in each cluster after the campaign has been running for three months will be enrolled together with their families. They will be identified through 3-monthly surveillance visits to all compounds identified at baseline; it is expected that recruitment will be achieved within a 6-month birth period. They will form the trial cohort and be followed 3-monthly until the end of the radio campaign. The intervention's impact on ECD nurturing care behaviours and ECD outcomes in the first 3 years of life will be evaluated.

DATA COLLECTION The trial will be supported by a surveillance system with regular 3-monthly visits by the cluster fieldworker (FW) to all households. These visits will be used to recruit the trial participants, maximize their follow-up during the trial and collect a variety of data on ECD behaviours and outcomes as well as process evaluation data on radio listening patterns. Details of all primary and secondary outcome assessments are presented in the next section.

SAMPLE SIZE Assessments are anticipated to be carried out on at least 100 children per cluster, after allowing for a maximum 20% loss to follow-up from recruitment. This will give 90% power to detect an effect size of 0.25, assuming an intra-class correlation of 0.01 (personal communication, from the Save the Children ECD trial in Rwanda) and 80% power to detect an effect size of 0.21. It will also give 90% power to detect an effect size of 0.4 on other ECD outcomes, the level achieved in several successful ECD interventions, assuming an intra-class correlation of 0.04, which is informed by unpublished results from the SPRING trial, and 80% power to detect an effect size of 0.33.

STATISTICAL METHODS Findings will be reported according to the CONSORT guidelines for cluster randomized trials. Analyses will be intention to treat and include all data from trial children and their families, regardless of their exposure to the radio campaign. Random-effects linear regression models using individual-level data will be used to adjust for the clustered design and any imbalances between intervention and control arms. Effect sizes will be presented as standardized mean differences with 95% confidence intervals (CI). The data analysis plan will be published prior to the end of recruitment.

PROCESS EVALUATION

Tracking and post-broadcast feedback

Independent radio trackers will determine if spots were broadcast as planned. Post-broadcast feedback on the campaign will be obtained through periodic focus group discussions (FGDs) and semi-structured key informant interviews. These data will be collected from at least two different communities every quarter, throughout the campaign duration.

Surveillance monitoring data

Monitoring data on radio coverage will be collected every 3 months from trial mothers including listenership in the past week and questions concerning child development advice heard on the radio. These data will also be collected from a separate monitoring cohort of mothers who participated in the baseline survey together with 6-monthly questions on key behaviours & knowledge targeted by the campaign.

QUALITATIVE RESEARCH Acceptability will be measured through 25-30 qualitative interviews with caregivers, who will be asked about their experience and views on the intervention approach and content. Data from the post-production feedback research will also be utilized. The mechanisms and barriers to behavioural uptake will be explored through qualitative interviews with a further sample of 25-30 families. Approximately five intervention communities will be selected to reflect the diversity within the study areas. Within communities' respondents will be selected to give diversity in key characteristics such as parity and socio-economic status.

Qualitative analysis will begin through the identification of themes during daily debriefing sessions. Key analytical categories will then be identified, and the interviews systematically indexed into the categories and interpreted and written up. During analysis, consensus coding methods will be used for initial interviews.

ECONOMIC EVALUATION

SUNRISE offers the opportunity to fully cost, from the provider perspective, a large-scale intervention to promote ECD. These provider costs will be used to calculate a range of incremental cost effectiveness ratios including cost per beneficiary and cost per unit of cognitive gain. The full provider costing will then form the basis for affordability estimates calculated as a percentage of national gross domestic product. The cost of a fully-scaled programme will also be compared with current health and education spending in context. Simple modelling of the gains from improved early childhood stimulation, using estimates from the Lancet Series in Early Child Development, would then be used to conduct a fiscal space analysis to explore the expansion in national income likely to arise from the effects of the program, and what percentage of that growth in income the program cost constitutes. Finally, the equity impact of this intervention will be measured, as early child development interventions are known to attenuate the effects of poverty.

DATA MANAGEMENT Data protection and confidentiality procedures will be specified and followed, in keeping with Good Clinical Practice (GCP) and the GDPR 2018. Data collection will be carried out using REDCap which is a secure web application for building and managing online surveys and databases; REDCap is 21 CFR Part 11, FISMA, HIPAA, and GDPR compliant. All data (including video observations) will be collected on secure, password protected handheld tablets within an encrypted database, with the data transferred daily to a secure password protected cloud server, managed by IPA in Ouagadougou. All electronic data will be backed up locally on a weekly basis on encrypted external hard drives and stored offsite in Ouagadougou. Encrypted transfer of pseudonymized quantitative data to LSHTM will take place monthly via secure internet connection to a GCP-compliant LSHTM database, which allows full auditing of all data input and edits. Qualitative interviews will be audio-recorded on digital audio recorders.

As video and audio data cannot be de-identified, transfer of this material to the UK will be done through UCL's Data Safe Haven, which is a dedicated highly secure system for storing and handling sensitive data. The Data Safe Haven has been certified to the ISO27001 information security standard and conforms to the NHS Information Governance Toolkit. Video recordings will be viewed only by members of the SUNRISE team and for the purposes of the research, unless further explicit written consent is obtained.

Data concerning cluster allocation will not be stored in the local or LSHTM research databases, but held separately by the trial statistician in a secure password protected file.

GOVERNANCE The trial will be overseen by an independent Trial Steering Committee (TSC) and Data Monitoring and Ethics Committtee (DMEC). TSC members are: Linda Richter (Chair), Jose Martines, Therese Stukel, Ali Sie. DMEC members are Rajiv Bahl (Chair)., Thierry Martens, Charlotte Tawiah-Agyemang, Susan Walker, Helen Weiss (independent statistician).

ETHICS APPROVAL As a non-CTIMP, no regulatory approvals for medicinal products will be required. The study will be reviewed by the ethics committees of the Ministry of Health, Burkina Faso, UCL and LSHTM. LSHTM will be the study sponsor. The trial will be registered with ClinicalTrials.gov prior to initiation.

ELIGIBILITY:
Inclusion Criteria:

* Live newborns with a birth date at least 3 months following the launch of the SUNRISE radio campaign will be eligible to be enrolled into the trial, together with their mothers.

Exclusion Criteria:

* Children with major infant congenital defects, children not living with their mother, and children with mothers who are not capable of participating in assessments.

For clarification:

* Age limits are for age at recruitment; children will be followed until age 30-32m.
* Early child development is the condition under study; this applies to all the participants. "Accepts Healthy Volunteers" is not meaningful in this trial.

Ages: 0 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1875 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Primary impact outcome: MDAT/GSED Child Development score | Assessed when child is age 30-32 months
  The Malawi Developmental Assessment Tool (MDAT) is a well validated developmental assessment, that has been designed and adapted to be appropriate in low resource settings and for a wide range of cultures and contexts. It consists of 136 test items, with 34 items covering gross and fine motor development, language and social development. A total score will be computed as an overall index of child development. The tool shows excellent inter-rater reliability and good sensitivity and specificity for identifying children with developmental disability/delays.
  Note: During the early phases of this trial, we will evaluate the evidence regarding the Global Scales of Early Development - Long Form (GSED-LF), which has more items than the MDAT and is expected to be a more sensitive assessment. Field testing of the GSED is nearly complete at the time of writing. If a decision is taken to use the GSED-LF this will be ratified by the TSC and approved by the REC.
Primary intermediate outcome: z-standardised observed sensitive responsiveness score using the National Institute of Child Health and Human Development (NICHD) sensitivity scales. | Assessed when child is age 8-20 months
  Sensitive responsiveness will be directly observed when the child is age 18-20m. Mothers will be video recorded carrying out a set of interactive tasks in which the child is introduced to a series of novel toys; this will last about 15 minutes. The videos will be independently coded, blind to whether the mother is in an intervention or control cluster, using the National Institute of Child Health and Human Development (NICHD) sensitivity scales, which assess "a parent's accuracy in perceiving and interpreting their infant's cues and their ability to react in a timely and appropriate manner".

SECONDARY OUTCOMES:
Secondary impact outcome: MDAT child development domain scores | Assessed when child is age 30-32 months
  The 4 MDAT developmental domain scores for gross and fine motor development, language and social development.
Secondary impact outcome: Five 6-monthly CREDI-LF total scores | Assessed 6-monthly, starting when the child is age 6-8 months until age 30-32 months.
  The long form of the Caregiver Reported Early Development Index (CREDI) is a developmental screening instrument designed specifically for large-scale surveys and evaluations for children aged zero to three years. It relies only on parental reporting and assesses 5 domains of early developmental milestones and behaviours, namely Motor, Language, Cognitive, Socio-Emotional and Mental Health, tailored to the child's age.
Secondary impact outcome: Five 6-monthly caregiver reported language development scores | Assessed 6-monthly, starting when the child is age 6-8 months until age 30-32 months.
  The Communicative Development Inventories (CDI) is one of the most widely used and well-validated tools for assessing early language development. The Words and Gestures short form (Level I) will be used for assessments up to including age 18-20m. This is a parent-reported checklist of early communication and receptive language, comprised of an 89-word vocabulary checklist with separate columns for comprehension and production. The Words and Sentences short form (Level II) of the CDI will be used at later ages. These measures contain a 100-word productive vocabulary checklist and a question about combining words.
Secondary intermediate outcome: The HOME-IT inventory (Home Observation for Measurement of the Environment, Infants & Toddler version) score | Assessed when the child is age 18-20 months.
  The HOME-IT inventory (Home Observation for Measurement of the Environment, Infants & Toddler version) provides a comprehensive assessment of the family environment, including the provision and variety of stimulating play materials, the organization of the physical environment, and levels of parental involvement, responsivity and acceptance of the child's behavior.
Secondary intermediate outcome: Five 6-monthly Family Care Indicators (FCI) scores. | Assessed 6-monthly, starting when the child is age 6-8 months until age 30-32 months.
  This will be based on the support for learning/stimulating environment section of the Family Care Indicators (FCI) survey, developed by UNICEF to assess key caregiving/family home environment variables considered critical for early child development. This has been used very extensively, including in the global MICS surveys.

OTHER OUTCOMES:
Tertiary outcome: Two Caregiver ECD Knowledge Scores | Assessed when the child is age 18-20 months and 30-32 months
  ECD knowledge will be assessed using a culturally adapted subset of questions from the Knowledge of Infant Development Inventory (KIDI). The KIDI measures factual knowledge of parental practices, child development processes and norms of behaviour for children 0-3 years of age. It is appropriate for use with persons of limited education and is considered to be culturally neutral.

CONTACTS AND LOCATIONS:
Overall Officials: Betty R Kirkwood, FMedSci, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Innovations for Poverty Action, Ouagadougou, Kadiogo, Burkina Faso

IPD SHARING:
Plan to Share IPD: Yes
The project will produce rich longitudinal data from trial recruitment in the first 6 months of life through to the follow-up at age 30-32 months. The data will be curated into a single anonymised STATA. sta file, including newly generated participant ID and cluster codes, variable labels, and defined missing values. All identifiable data or data that may risk de-anonymisation (such as DOBs, personal names or cluster and village names) will be removed. Alongside the main study data file, codebooks and a detailed dataset guide will be produced to support correct and efficient data usage. Derived and computed variables and processing steps will be made available through annotated STATA analysis .do scripts.
  Videos and qualitative interview data, where anonymization is either not possible or there is a high risk of individuals being identified, will not be made publicly available. Suitably qualified researchers will be able to access these data under strict collaboration agreements.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 3 years from study completion, which is anticipated to be October 2025
Access Criteria: TBC

REFERENCES:
- [Background] Black MM, Walker SP, Fernald LCH, Andersen CT, DiGirolamo AM, Lu C, McCoy DC, Fink G, Shawar YR, Shiffman J, Devercelli AE, Wodon QT, Vargas-Baron E, Grantham-McGregor S; Lancet Early Childhood Development Series Steering Committee. Early childhood development coming of age: science through the life course. Lancet. 2017 Jan 7;389(10064):77-90. doi: 10.1016/S0140-6736(16)31389-7. Epub 2016 Oct 4. PMID 27717614
- [Background] Richter LM, Daelmans B, Lombardi J, Heymann J, Boo FL, Behrman JR, Lu C, Lucas JE, Perez-Escamilla R, Dua T, Bhutta ZA, Stenberg K, Gertler P, Darmstadt GL; Paper 3 Working Group and the Lancet Early Childhood Development Series Steering Committee. Investing in the foundation of sustainable development: pathways to scale up for early childhood development. Lancet. 2017 Jan 7;389(10064):103-118. doi: 10.1016/S0140-6736(16)31698-1. Epub 2016 Oct 4. PMID 27717610
- [Background] McCoy DC, Sudfeld CR, Bellinger DC, Muhihi A, Ashery G, Weary TE, Fawzi W, Fink G. Development and validation of an early childhood development scale for use in low-resourced settings. Popul Health Metr. 2017 Feb 9;15(1):3. doi: 10.1186/s12963-017-0122-8. PMID 28183307
- [Background] Kariger P, Frongillo EA, Engle P, Britto PM, Sywulka SM, Menon P. Indicators of family care for development for use in multicountry surveys. J Health Popul Nutr. 2012 Dec;30(4):472-86. doi: 10.3329/jhpn.v30i4.13417. PMID 23304914
- [Background] Gladstone M, Lancaster GA, Umar E, Nyirenda M, Kayira E, van den Broek NR, Smyth RL. The Malawi Developmental Assessment Tool (MDAT): the creation, validation, and reliability of a tool to assess child development in rural African settings. PLoS Med. 2010 May 25;7(5):e1000273. doi: 10.1371/journal.pmed.1000273. PMID 20520849
- [Derived] Palmer T, Clare A, Fearon P, Head R, Hill Z, Kagone B, Kirkwood B, Manu A, Skordis J; SUNRISE team. Cost-effectiveness of a radio intervention to stimulate early childhood development: protocol for an economic evaluation of the SUNRISE trial in Burkina Faso. BMJ Open. 2024 Apr 16;14(4):e080905. doi: 10.1136/bmjopen-2023-080905. PMID 38626956
- [Derived] Dumbaugh M, Belem M, Kousse S, Ouoba P, Sankoudouma A, Tchibozo AM, Fearon P, Hollowell J, Hill Z; SUNRISE team. 'Children awaken by playing': a qualitative exploration of caregivers' norms, beliefs and practices related to young children's learning and early childhood development in rural Burkina Faso. BMJ Open. 2023 Oct 29;13(10):e075675. doi: 10.1136/bmjopen-2023-075675. PMID 37899153

DOCUMENTS (2):
  • Study Protocol (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT05335395/Prot_000.pdf
  • Informed Consent Form (2022-01-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT05335395/ICF_001.pdf